CLINICAL TRIAL: NCT03754036
Title: Effect of Increasing Sleep Duration on Insulin Sensitivity in Adolescents Having Risk Factors for Type 2 Diabetes
Brief Title: Sleep Extension and Insulin Sensitivity in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Jean-Philippe Chaput, Research Scientist, Children's Hospital of Eastern Ontario Research Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 17/63X
Record Dates: First submitted 2018-11-23; First posted 2018-11-27 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Sleep

STUDY DESIGN:
Intervention Model Description: Sleep restriction (-1.5 hours of sleep per day for 1 week) and Sleep extension (+1.5 hours of sleep per day for 1 week)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Extension (Experimental): Increase in time in bed of 1.5 hours per night for one week
  Interventions: Behavioral: Sleep manipulation
- Sleep Restriction (Experimental): Decrease in time in bed of 1.5 hours per night for one week
  Interventions: Behavioral: Sleep manipulation

INTERVENTIONS:
Behavioral: Sleep manipulation — Participants will sleep their typical amount at home for 1 week and will then be randomized to either increase or decrease their time in bed by 1.5 hours per night for 1 week, completing the alternate schedule on the fourth week (washout period of 1 week between sleep conditions). This procedure will result in a targeted 3-hour time in bed difference between conditions. Sleep will be objectively measured using actigraphy (Actiwatch) and sleep schedule adherence will be promoted by providing fixed bedtimes and wake times during the experimental weeks, and will be monitored through phone calls to the research center.

SUMMARY:
BACKGROUND: The influence of sleep extension on glucose homeostasis in adolescents at risk for type 2 diabetes is unknown. This issue is of high clinical relevance given the high prevalence of sleep deprivation in this population and the accumulating body of evidence indicating that having a good night's sleep is important for the prevention of chronic diseases including type 2 diabetes.

OBJECTIVE: To determine if extending sleep duration improves insulin sensitivity in adolescents presenting with risk factors for type 2 diabetes.

HYPOTHESIS: It was hypothesized that compared with decreasing sleep duration, increasing sleep duration by 1.5 hours over 1 week will improve insulin sensitivity.

METHODS: Using a randomized, counterbalanced, 2-condition crossover design, 30 obese adolescents between 13 and 18 years of age who have insulin resistance will complete the study. Participants will sleep their typical amount at home for 1 week and will then be randomized to either increase or decrease their time in bed by 1.5 hours per night for 1 week, completing the alternate schedule on the fourth week (washout period of at least 1 week between sleep conditions). This procedure will result in a targeted 3-hour time in bed difference between conditions. Sleep will be objectively measured using actigraphy (Actiwatch) and sleep schedule adherence will be promoted by providing fixed bedtimes and wake times during the experimental weeks, and will be monitored through phone calls to the research center. Participants will also be compensated for keeping the sleep schedule and daily calls to enhance adherence. The outcome measures will then be compared between both sleep conditions at the end (on day 8 of each study week). The primary outcome measure will be insulin sensitivity as measured by the Matsuda index (total body insulin sensitivity). Secondary outcomes will include the homeostasis model assessment of insulin resistance (HOMA-IR), blood lipids, food intake and physical activity. Repeated measures analysis using the mixed model will be used to assess the effect of the two sleep interventions on insulin sensitivity.

RELEVANCE: The study will provide the first robust clinical evidence to determine if increasing sleep duration in youth at risk for type 2 diabetes improves insulin sensitivity. This information will be essential for clinical and public health guidelines for type 2 diabetes prevention among adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents between the ages of 13 and 18 with obesity (body mass index greater than the 95th percentile) and dyslipidemia (total cholesterol ≥ 200 mg/dL; low-density lipoprotein cholesterol ≥ 130 mg/dL; non-high-density lipoprotein ≥ 145 mg/dL; triglycerides ≥ 130 mg/dL; and high-density lipoprotein < 40 mg/dL)
* Adolescents who report between 6.5-8 hours of sleep per night will be eligible to ensure that adolescents can extend and restrict sleep duration without reaching a ceiling for what can be achieved (i.e. 8-10 hours/night of sleep is recommended at this age) while limiting excessive sleep deprivation

Exclusion Criteria:

* History of a chronic medical or psychiatric condition
* Use of medications that could affect sleep or glucose homeostasis (e.g., metformin, thyroid medication, stimulant medication, etc.)
* History of sleep problems (e.g. sleep apnea).

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2021-12-12 (Actual)

PRIMARY OUTCOMES:
Insulin sensitivity | On day 8 of each sleep condition (2 time points)
  Assessed by the Matsuda index during a 2-hour oral glucose tolerance test (OGTT)

SECONDARY OUTCOMES:
Insulin sensitivity | On day 8 of each sleep condition (2 time points)
  HOMA-IR
Blood lipids | On day 8 of each sleep condition (2 time points)
  HDL-cholesterol, LDL-cholesterol, triglycerides, total cholesterol
Food intake | On days 5, 6 and 7 of each sleep condition (2 time points)
  3-day dietary record
Physical activity level | During each 7-day sleep condition (2 time points)
  Minutes per day of moderate-to-vigorous physical activity as assessed by accelerometry

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital of Eastern Ontario Research Institute, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dutil C, Podinic I, Featherstone RB, Eaton A, Sadler CM, Goldfield GS, Hadjiyannakis S, Gruber R, Tremblay MS, Prud'homme D, Chaput JP. Sleep and insulin sensitivity in adolescents at risk of type 2 diabetes: the Sleep Manipulation in Adolescents at Risk of Type 2 Diabetes randomized crossover study. Sleep. 2024 May 10;47(5):zsad313. doi: 10.1093/sleep/zsad313. PMID 38070132